CLINICAL TRIAL: NCT04942743
Title: Clinical & MRI Finding of TMJ Disk Perforation
Status: Completed | Type: Observational
Sponsor: Al-Azhar University (Other)
Responsible Party: Principal Investigator, Ayman Hegab, associate professor of oral and maxillofacial surgery, Al-Azhar University
Other Study IDs: AUAREC20200501-12
Record Dates: First submitted 2021-06-24; First posted 2021-06-28 (Actual); Last update posted 2021-07-01 (Actual); Status verified 2021-06

CONDITIONS: TMJ Disc Disorder

STUDY DESIGN:
Observational Model: Other | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- control group: patients with normal TMJ
  Interventions: Diagnostic Test: MRI
- Study group: patients with TMJ internal derangement
  Interventions: Diagnostic Test: MRI

INTERVENTIONS:
Diagnostic Test: MRI — MRI OF TMJ

SUMMARY:
the study aimed to evaluate the clinical and MRI finding of TMJ with disk perforation with predication of the risk factors.

DETAILED DESCRIPTION:
The retrospective study included patients seeking treatment for TMD at Al-Azhar University Hospital and the outpatient clinic at the Faculty of Dental Medicine of Al-Azahr University. The sample originally included patients who provided consent to participate in this study and who ultimately underwent treatment for TMJD between 2008 and 2019.

Exclusion Inclusion criteria: Patients were included if they were older than 18 years and diagnosed with TMJD. criteria for this study included systemic diseases (the presence of polyarthritis or other rheumatic diseases), contraindications for MRI (e.g., implanted metal or medical devices, claustrophobia), the presence of neurologic disorders, head and neck cancer, oral submucous ﬁbrosis, a history of TMJ surgery, a history of previous nonsurgical treatment such as occlusal splints, and a history of joint injection with HA/PRP. Trauma patients with subcondylar fracture and patients with congenital and developmental disorders of the TMJ were also excluded from the study.

the study included 2 groups group 1: normal TMJ patients group 2: patients with TMJ internal derangement

ELIGIBILITY:
Inclusion Criteria:

* patients seeking treatment for TMD at Al-Azhar University Hospital and the outpatient clinic at the Faculty of Dental Medicine of Al-Azahr University.

Exclusion Criteria:

* Patients were included if they were older than 18 years and diagnosed with TMJD. criteria for this study included systemic diseases (the presence of polyarthritis or other rheumatic diseases), contraindications for MRI (e.g., implanted metal or medical devices, claustrophobia), the presence of neurologic disorders, head and neck cancer, oral submucous ﬁbrosis, a history of TMJ surgery, a history of previous nonsurgical treatment such as occlusal splints, and a history of joint injection with HA/PRP. Trauma patients with subcondylar fracture and patients with congenital and developmental disorders of the TMJ were also excluded from the study.

Ages: 19 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: The sample originally included patients who provided consent to participate in this study and who ultimately underwent treatment for TMJD between 2008 and 2019.
Sampling Method: Non-Probability Sample
Enrollment: 900 (Actual)
Dates: Start 2020-01-12 (Actual); Primary Completion 2020-12-31 (Actual); Study Completion 2021-06-15 (Actual)

PRIMARY OUTCOMES:
joint pain (VAS), | pre treatment
  pain index scores were measured using a 10-point visual analogue scale (VAS), with 0 indicating absence of pain and 10 indicating the worst pain.
(MVMO) | pretreatment
  mouth opening

SECONDARY OUTCOMES:
joint sound | pretreatment
  joint sound was then determined by combining 3 means: (1) palpation of the TMJ zone by the clinician, (2) the patient's self-reporting regarding whether the joint sound could be heard, and (3) auscultation of the TMJ zone with the stethoscope.

CONTACTS AND LOCATIONS:
Overall Officials: Ayman Hegab, Phd, Principal Investigator — Al-Azhar University
Locations (1):
- Faculty of Dental Medicine Alazhar University, Cairo, Nasr City, Egypt

IPD SHARING:
Plan to Share IPD: No